CLINICAL TRIAL: NCT02573727
Title: ''To Compare the Response Rate of Noradrenaline vs. Terlipressin in Hepatorenal Syndrome in Patients With Acute on Chronic Liver Failure'
Brief Title: To Compare the Response Rate of Noradrenaline vs. Terlipressin in Hepatorenal Syndrome in Patients With Acute on Chronic Liver Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-004
Record Dates: First submitted 2015-10-05; First posted 2015-10-12 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2016-07

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Norepinephrine; Albumins; Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nor Adrenaline + Albumin (Experimental): Intravenous continous infusion of terlipressin at the dose of 2 mg every 24 hours with the maximum daily cumulative dose of 12 mg/day.
  In case of no response the dose of the terlipressin will be progressively increased to the maximum infusion dose of 12 mg/24 hour.
  Patients will be given 1g/Kg of albumin per day, which will be discontinued if CVP is more than 18 cm H2O.
  Interventions: Drug: Nor adrenaline + albumin
- Terlipressin + Albumin (Active Comparator): Continuous IV infusion of NA starting at 0.5 mg/h with doubling of dose after every 4 hours designed to achieve an increase in MAP of at least 10 mmHg or an increase in 4-h urine output of more than 200 ml. When one of these goals was not achieved, the noradrenaline dose was increased every 4 h in steps of 0.5 mg/h, up to the maximum dose of 3 mg/h.
  Patients will be given 1g/Kg of albumin per day, which will be discontinued if CVP is more than 18 cm H2O.
  Interventions: Drug: Terlipressin + albumin

INTERVENTIONS:
Drug: Nor adrenaline + albumin
  Arms: Nor Adrenaline + Albumin
Drug: Terlipressin + albumin
  Arms: Terlipressin + Albumin

SUMMARY:
Continous infusion of nor adrenaline + albumin Continous infusion of terlipressin + albumin Response will assessed at every 48 hour (i) Complete response: Regression of acute kidney injury stage with reduction of S. Cr within 0.3 mg/dl of baseline (ii) Partial response: Regression of acute kidney injury stage with reduction of S. Cr to ≥0.3 mg/dl above baseline (iii) No response: No regression of acute kidney injury

Treatment will be extended until reversal of HRS (decrease in creatinine below 1.5 mg/dL) or for a maximum of 7 days after rescue treatment will be followed.

If intolerant to terlipressin, excluded from study and rescue treatment will be given in form of noradrenaline or octreotide and midodrine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute on chronic liver failure presenting with hepatorenal syndrome
2. Patients consented for the study protocol by signing the informed consent.

Exclusion Criteria:

1. Age less than 18 years
2. Decompensated cirrhotics
3. Evidence of chronic kidney disease
4. Patients undergoing renal replacement therapy (hemo-dialysis/renal transplantation).
5. Post liver transplantation patients.
6. History of coronary artery disease, ischaemic cardiomyopathy, ventricular arrhythmia, or peripheral vascular disease.
7. Patients with obstructive uropathy.
8. Patient who withdrew or non complaint to the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Response to treatment in each intervention group | 14 days
  Complete response: Regression of acute kidney injury stage with reduction of S. Cr within 0.3 mg/dl of baseline (ii) Partial response: Regression of acute kidney injury stage with reduction of S. Cr to ≥0.3 mg/dl above baseline (iii) No response: No regression of acute kidney injury.

SECONDARY OUTCOMES:
Survival | 28 days
Drug related Side effects/complications | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Vinod Arora, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India